CLINICAL TRIAL: NCT02628873
Title: Can Contrast Infused Sonography Using Air Bubbles Replace Hysterosalpingogram as the Diagnostic Evaluation of Fallopian Tube Patency Following Hysteroscopic Sterilization Using Essure
Brief Title: Can SIS Using Air Bubbles Replace HSG for Fallopian Tubal Patency After Essure Placement
Acronym: HyCoSy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Essure no longer sold in the US after Dec 2018; Sponsor requested trial be ended
Sponsor: Wright State University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: Lindheim2015-01
Record Dates: First submitted 2015-10-05; First posted 2015-12-11 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Contraception
Keywords: HSG; HyCoSy; Contraception; Essure; Saline Infused sonography; SIS; Air bubbles

STUDY DESIGN:
Intervention Model Description: Cross over study in which participants receive one diagnostic test (SSI or HSG), then receive the other.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor does not know which procedure was received first or second.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm 1 (HyCoSy followed by HSG) (Experimental): HyCoSy procedure followed by HSG procedure
  Interventions: Device: HyCoSy
- Arm 2 (HSG followed by HyCoSy) (Experimental): HSG procedure followed by HyCoSy procedure
  Interventions: Device: HyCoSy

INTERVENTIONS:
Device: HyCoSy — Saline infused sonogram in which air bubbles are delivered via the FemVue saline air device in order to evaluate the patency (openness) of the fallopian tubes
  Other Names: Fem Vue; Saline Air Device; Saline infused sonogram

SUMMARY:
The study evaluates whether saline infused sonography (SIS) with directed air bubbles for hysterosalpingo-contrast sonography (HyCoSy) is as good as or better than X-ray hysterosalpingography (HSG) for determining whether fallopian tubes are open or closed in patients who are undergoing an Essure confirmation test.

DETAILED DESCRIPTION:
The gold standard for evaluating whether fallopian tubes are open versus closed is the X-ray hysterosalpingography (HSG). HSG is a radiologic procedure that is performed to verify that placement of the Essure tubal ligation inserts have successfully blocked the fallopian tubes. However, this procedure involved exposure to radiation. The saline infused sonography (SIS) with directed air bubbles for hysterosalpingo-contrast sonography (HyCoSy) does not involve radiation and can be done in a physician's office. The HyCoSy air bubble device may be a lower cost, safer alternative procedure if it can be shown to provide similar results for tubal patency.

This study will compare the HyCoSy procedure results with the HSG procedure results in women who require the HSG procedure after receiving Essure tubal ligation inserts for their Essure confirmation test.

Women will be randomized to receive the HycoSy procedure first, followed by the HSG procedure or to the reverse order. Two independent readers will review the video results for both procedures to determine the degree of agreement on tubal patency.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of normal Pap smear within 1 year prior to enrollment into study.
* Written informed consent given
* Need for evaluation of tubal status for post-Essure tubal occlusion
* Negative urine pregnancy test

Exclusion Criteria:

* History of unresolved dysfunctional uterine bleeding (DUB).
* History of a hysterectomy.
* Current urogenital disease.
* History of allergic response to IVP dye (exclusion for HSG).
* Abnormal pap smear.
* Positive urine pregnancy test.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lindheim, MD, Principal Investigator — Wright State University
Locations (1):
- Wright State Physicians, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share date due to small sample size

REFERENCES:
- [Background] Smith RD. Contemporary hysteroscopic methods for female sterilization. Int J Gynaecol Obstet. 2010 Jan;108(1):79-84. doi: 10.1016/j.ijgo.2009.07.026. PMID 19716128
- [Background] Practice Committee of the American Society for Reproductive Medicine. Optimal evaluation of the infertile female. Fertil Steril. 2006 Nov;86(5 Suppl 1):S264-7. doi: 10.1016/j.fertnstert.2006.08.041. No abstract available. PMID 17055838
- [Background] Radic V, Canic T, Valetic J, Duic Z. Advantages and disadvantages of hysterosonosalpingography in the assessment of the reproductive status of uterine cavity and fallopian tubes. Eur J Radiol. 2005 Feb;53(2):268-73. doi: 10.1016/j.ejrad.2004.02.015. PMID 15664291
- [Background] Veersema S, Vleugels MP, Moolenaar LM, Janssen CA, Brolmann HA. Unintended pregnancies after Essure sterilization in the Netherlands. Fertil Steril. 2010 Jan;93(1):35-8. doi: 10.1016/j.fertnstert.2008.10.005. Epub 2008 Nov 21. PMID 19027109
- [Background] The American Fertility Society classifications of adnexal adhesions, distal tubal occlusion, tubal occlusion secondary to tubal ligation, tubal pregnancies, mullerian anomalies and intrauterine adhesions. Fertil Steril. 1988 Jun;49(6):944-55. doi: 10.1016/s0015-0282(16)59942-7. No abstract available. PMID 3371491
- [Background] Okonofua FE, Essen UI, Nimalaraj T. Hysterosalpingography versus laparoscopy in tubal infertility: comparison based on findings at laparatomy. Int J Gynaecol Obstet. 1989 Feb;28(2):143-7. doi: 10.1016/0020-7292(89)90474-8. PMID 2563701
- [Background] Musich JR, Behrman SJ. Infertility laparoscopy in perspective: review of five hundred cases. Am J Obstet Gynecol. 1982 Jun 1;143(3):293-303. doi: 10.1016/0002-9378(82)90818-3. PMID 6211097
- [Background] al-Badawi IA, Fluker MR, Bebbington MW. Diagnostic laparoscopy in infertile women with normal hysterosalpingograms. J Reprod Med. 1999 Nov;44(11):953-7. PMID 10589406
- [Background] Romano F, Cicinelli E, Anastasio PS, Epifani S, Fanelli F, Galantino P. Sonohysterography versus hysteroscopy for diagnosing endouterine abnormalities in fertile women. Int J Gynaecol Obstet. 1994 Jun;45(3):253-60. doi: 10.1016/0020-7292(94)90251-8. PMID 7926245
- [Background] Nannini R, Chelo E, Branconi F, Tantini C, Scarselli GF. Dynamic echohysteroscopy: a new diagnostic technique in the study of female infertility. Acta Eur Fertil. 1981 Jun;12(2):165-71. No abstract available. PMID 7293673
- [Background] Parsons AK, Lense JJ. Sonohysterography for endometrial abnormalities: preliminary results. J Clin Ultrasound. 1993 Feb;21(2):87-95. doi: 10.1002/jcu.1870210203. PMID 8381140
- [Background] Lindheim SR, Adsuar N, Kushner DM, Pritts EA, Olive DL. Sonohysterography: a valuable tool in evaluating the female pelvis. Obstet Gynecol Surv. 2003 Nov;58(11):770-84. doi: 10.1097/01.OGX.0000094386.63363.D7. PMID 14581828
- [Background] Mitri FF, Andronikou AD, Perpinyal S, Hofmeyr GJ, Sonnendecker EW. A clinical comparison of sonographic hydrotubation and hysterosalpingography. Br J Obstet Gynaecol. 1991 Oct;98(10):1031-6. doi: 10.1111/j.1471-0528.1991.tb15342.x. PMID 1751435
- [Background] Richman TS, Viscomi GN, deCherney A, Polan ML, Alcebo LO. Fallopian tubal patency assessed by ultrasound following fluid injection. Work in progress. Radiology. 1984 Aug;152(2):507-10. doi: 10.1148/radiology.152.2.6539931.
- [Background] Session DR, Lerner JP, Tchen CK, Kelly AC. Ultrasound-guided fallopian tube cannulation using Albunex. Fertil Steril. 1997 May;67(5):972-4. doi: 10.1016/s0015-0282(97)81420-3. PMID 9130913
- [Background] Campbell S, Bourne TH, Tan SL, Collins WP. Hysterosalpingo contrast sonography (HyCoSy) and its future role within the investigation of infertility in Europe. Ultrasound Obstet Gynecol. 1994 May 1;4(3):245-53. doi: 10.1046/j.1469-0705.1994.04030245.x. PMID 12797192
- [Background] Luciano DE, Exacoustos C, Johns DA, Luciano AA. Can hysterosalpingo-contrast sonography replace hysterosalpingography in confirming tubal blockage after hysteroscopic sterilization and in the evaluation of the uterus and tubes in infertile patients? Am J Obstet Gynecol. 2011 Jan;204(1):79.e1-5. doi: 10.1016/j.ajog.2010.08.065. PMID 21187197
- [Background] Emanuel MH, van Vliet M, Weber M, Exalto N. First experiences with hysterosalpingo-foam sonography (HyFoSy) for office tubal patency testing. Hum Reprod. 2012 Jan;27(1):114-7. doi: 10.1093/humrep/der367. Epub 2011 Nov 6. PMID 22064649
- [Background] Holz K, Becker R, Schurmann R. Ultrasound in the investigation of tubal patency. A meta-analysis of three comparative studies of Echovist-200 including 1007 women. Zentralbl Gynakol. 1997;119(8):366-73. PMID 9286072
- [Background] Andersen AN, Yue Z, Meng FJ, Petersen K. Low implantation rate after in-vitro fertilization in patients with hydrosalpinges diagnosed by ultrasonography. Hum Reprod. 1994 Oct;9(10):1935-8. doi: 10.1093/oxfordjournals.humrep.a138362. PMID 7844229
- [Background] Strandell A, Bourne T, Bergh C, Granberg S, Asztely M, Thorburn J. The assessment of endometrial pathology and tubal patency: a comparison between the use of ultrasonography and X-ray hysterosalpingography for the investigation of infertility patients. Ultrasound Obstet Gynecol. 1999 Sep;14(3):200-4. doi: 10.1046/j.1469-0705.1999.14030200.x. PMID 10550881
- [Background] Stumpf PG, March CM. Febrile morbidity following hysterosalpingography: identification of risk factors and recommendations for prophylaxis. Fertil Steril. 1980 May;33(5):487-92. doi: 10.1016/s0015-0282(16)44712-6. PMID 7371880
- [Background] Moore DE, Segars JH Jr, Winfield AC, Page DL, Eisenberg AD, Holburn GE. Effects of contrast agents on the fallopian tube in a rabbit model. Radiology. 1990 Sep;176(3):721-4. doi: 10.1148/radiology.176.3.2167499.
- [Background] Thurmond AS, Hedgpeth PL, Scanlan RM. Selective injection of contrast media: inflammatory effects on rabbit fallopian tubes. Radiology. 1991 Jul;180(1):97-9. doi: 10.1148/radiology.180.1.1647040.
- [Background] Lindequist S, Justesen P, Larsen C, Rasmussen F. Diagnostic quality and complications of hysterosalpingography: oil- versus water-soluble contrast media--a randomized prospective study. Radiology. 1991 Apr;179(1):69-74. doi: 10.1148/radiology.179.1.1848715.
- [Background] Acton CM, Devitt JM, Ryan EA. Hysterosalpingography in infertility--an experience of 3,631 examinations. Aust N Z J Obstet Gynaecol. 1988 May;28(2):127-33. doi: 10.1111/j.1479-828x.1988.tb01641.x. No abstract available. PMID 2976272
- [Background] Mohiyiddeen L, Hardiman A, Fitzgerald C, Hughes E, Mol BW, Johnson N, Watson A. Tubal flushing for subfertility. Cochrane Database Syst Rev. 2015 May 1;2015(5):CD003718. doi: 10.1002/14651858.CD003718.pub4. PMID 25929235
- [Background] Boyer P, Territo MC, de Ziegler D, Meldrum DR. Ethiodol inhibits phagocytosis by pelvic peritoneal macrophages. Fertil Steril. 1986 Oct;46(4):715-7. doi: 10.1016/s0015-0282(16)49657-3. No abstract available. PMID 3019786
- [Background] Johnson JV, Montoya IA, Olive DL. Ethiodol oil contrast medium inhibits macrophage phagocytosis and adherence by altering membrane electronegativity and microviscosity. Fertil Steril. 1992 Sep;58(3):511-7. doi: 10.1016/s0015-0282(16)55254-6. PMID 1325928
- [Background] Darby SC, Wall BF. The genetically significant dose from diagnostic radiology in Great Britain. Radiography. 1981 Sep;47(561):200-2. No abstract available. PMID 7330172
- [Background] Karande VC, Pratt DE, Balin MS, Levrant SG, Morris RS, Gleicher N. What is the radiation exposure to patients during a gynecoradiologic procedure? Fertil Steril. 1997 Feb;67(2):401-3. doi: 10.1016/S0015-0282(97)81931-0. PMID 9022623
- [Background] Volpi E, Zuccaro G, Patriarca A, Rustichelli S, Sismondi P. Transvaginal sonographic tubal patency testing using air and saline solution as contrast media in a routine infertility clinic setting. Ultrasound Obstet Gynecol. 1996 Jan;7(1):43-8. doi: 10.1046/j.1469-0705.1996.07010043.x. PMID 8932631
- [Background] Swart P, Mol BW, van der Veen F, van Beurden M, Redekop WK, Bossuyt PM. The accuracy of hysterosalpingography in the diagnosis of tubal pathology: a meta-analysis. Fertil Steril. 1995 Sep;64(3):486-91. doi: 10.1016/s0015-0282(16)57781-4. PMID 7641899
- [Background] Sulak PJ, Letterie GS, Coddington CC, Hayslip CC, Woodward JE, Klein TA. Histology of proximal tubal occlusion. Fertil Steril. 1987 Sep;48(3):437-40. PMID 2957237
- [Background] Hamed HO, Shahin AY, Elsamman AM. Hysterosalpingo-contrast sonography versus radiographic hysterosalpingography in the evaluation of tubal patency. Int J Gynaecol Obstet. 2009 Jun;105(3):215-7. doi: 10.1016/j.ijgo.2009.02.001. Epub 2009 Mar 31. PMID 19339010
- [Background] Chenia F, Hofmeyr GJ, Moolla S, Oratis P. Sonographic hydrotubation using agitated saline: a new technique for improving fallopian tube visualization. Br J Radiol. 1997 Aug;70(836):833-6. doi: 10.1259/bjr.70.836.9486049.
- [Background] Exacoustos C, Zupi E, Carusotti C, Lanzi G, Marconi D, Arduini D. Hysterosalpingo-contrast sonography compared with hysterosalpingography and laparoscopic dye pertubation to evaluate tubal patency. J Am Assoc Gynecol Laparosc. 2003 Aug;10(3):367-72. doi: 10.1016/s1074-3804(05)60264-2. PMID 14567814
- [Background] Kiyokawa K, Masuda H, Fuyuki T, Koseki M, Uchida N, Fukuda T, Amemiya K, Shouka K, Suzuki K. Three-dimensional hysterosalpingo-contrast sonography (3D-HyCoSy) as an outpatient procedure to assess infertile women: a pilot study. Ultrasound Obstet Gynecol. 2000 Dec;16(7):648-54. doi: 10.1046/j.1469-0705.2000.00327.x. PMID 11169373
- [Background] Deichert U, Schleif R, van de Sandt M, Juhnke I. Transvaginal hysterosalpingo-contrast-sonography (Hy-Co-Sy) compared with conventional tubal diagnostics. Hum Reprod. 1989 May;4(4):418-24. doi: 10.1093/oxfordjournals.humrep.a136920. PMID 2526153
- [Background] Degenhardt F, Jibril S, Eisenhauer B. Hysterosalpingo-contrast sonography (HyCoSy) for determining tubal patency. Clin Radiol. 1996 Feb;51 Suppl 1:15-8. No abstract available. PMID 8605765
- [Background] Patel MD, Acord DL, Young SW. Likelihood ratio of sonographic findings in discriminating hydrosalpinx from other adnexal masses. AJR Am J Roentgenol. 2006 Apr;186(4):1033-8. doi: 10.2214/AJR.05.0091. PMID 16554575
- [Background] Reis MM, Soares SR, Cancado ML, Camargos AF. Hysterosalpingo contrast sonography (HyCoSy) with SH U 454 (Echovist) for the assessment of tubal patency. Hum Reprod. 1998 Nov;13(11):3049-52. doi: 10.1093/humrep/13.11.3049. PMID 9853854
- [Background] Tanawattanacharoen S, Suwajanakorn S, Uerpairojkit B, Boonkasemsanti W, Virutamasen P. Transvaginal hysterosalpingo-contrast sonography (HyCoSy) compared with chromolaparoscopy. J Obstet Gynaecol Res. 2000 Feb;26(1):71-5. doi: 10.1111/j.1447-0756.2000.tb01205.x. PMID 10761336
- [Background] Shi WT, Forsberg F, Bautista R, Vecchio C, Bernardi R, Goldberg BB. Image enhancement by acoustic conditioning of ultrasound contrast agents. Ultrasound Med Biol. 2004 Feb;30(2):191-8. doi: 10.1016/j.ultrasmedbio.2003.10.007. PMID 14998671
- [Background] Connor V. Contrast infusion sonography in the post-Essure setting. J Minim Invasive Gynecol. 2008 Jan-Feb;15(1):56-61. doi: 10.1016/j.jmig.2007.07.008. PMID 18262145
- [Background] Hurd WW, Wyckoff ET, Reynolds DB, Amesse LS, Gruber JS, Horowitz GM. Patient rotation and resolution of unilateral cornual obstruction during hysterosalpingography. Obstet Gynecol. 2003 Jun;101(6):1275-8. doi: 10.1016/s0029-7844(03)00361-2. PMID 12798536
- [Background] Kurt M, Shaikh KA, Peterson L, Kurrelmeyer KM, Shah G, Nagueh SF, Fromm R, Quinones MA, Zoghbi WA. Impact of contrast echocardiography on evaluation of ventricular function and clinical management in a large prospective cohort. J Am Coll Cardiol. 2009 Mar 3;53(9):802-10. doi: 10.1016/j.jacc.2009.01.005. PMID 19245974
- [Background] Hamilton JA, Larson AJ, Lower AM, Hasnain S, Grudzinskas JG. Evaluation of the performance of hysterosalpingo contrast sonography in 500 consecutive, unselected, infertile women. Hum Reprod. 1998 Jun;13(6):1519-26. doi: 10.1093/humrep/13.6.1519. PMID 9688385
- [Background] Lanzani C, Savasi V, Leone FPG, Ratti M, Ferrazzi E. Two-dimensional HyCoSy with contrast tuned imaging technology and a second-generation contrast media for the assessment of tubal patency in an infertility program. Fertil Steril. 2009 Sep;92(3):1158-1161. doi: 10.1016/j.fertnstert.2008.07.1746. Epub 2008 Oct 1. PMID 18829020
- [Background] Jeanty P, Besnard S, Arnold A, Turner C, Crum P. Air-contrast sonohysterography as a first step assessment of tubal patency. J Ultrasound Med. 2000 Aug;19(8):519-27. doi: 10.7863/jum.2000.19.8.519. PMID 10944037
- [Result] Luong E, Ludwin A, Winter T, Yaklic J, Maxwell RA, Bhagavath B, Lindheim SR. Saline-Air Hysterosalpingo-Contrast Sonography Is Equivalent to the Modified Hysterosalpingogram Following Hysteroscopic Sterilization. Ultrasound Q. 2020 Jun;36(2):138-145. doi: 10.1097/RUQ.0000000000000488. PMID 32511207

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from existing practice and clinic patients who had the Essure device placed for contraception.
Groups:
- Arm 1 (HyCoSy Followed by HSG): HyCoSy followed by HSG
  HyCoSy: Saline infused sonogram in which air bubbles are delivered via the FemVue saline air device in order to evaluate the patency (openness) of the fallopian tubes
- Arm 2 (HSG Followed by HyCoSy): HSG followed by HyCoSy
  HyCoSy: Saline infused sonogram in which air bubbles are delivered via the FemVue saline air device in order to evaluate the patency (openness) of the fallopian tubes
Period: First Test (1 Hour)
Arm/Group | Arm 1 (HyCoSy Followed by HSG) | Arm 2 (HSG Followed by HyCoSy)
Started | 14 | 7
Completed | 14 | 7
Not Completed | 0 | 0
Period: Break (1 Hour)
Arm/Group | Arm 1 (HyCoSy Followed by HSG) | Arm 2 (HSG Followed by HyCoSy)
Started | 14 | 7
Completed | 14 | 6
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Test (1 Hour)
Arm/Group | Arm 1 (HyCoSy Followed by HSG) | Arm 2 (HSG Followed by HyCoSy)
Started | 14 | 6
Completed | 13 | 6
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Number of participants are those who completed all assessments.
  Units of analysis for evaluation of the diagnostic tests is # fallopian tubes (open versus closed). All participants had 2 fallopian tubes.
Units Other Than Participants: # fallopian tubes
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (HyCoSy Followed by HSG) | Arm 2 (HSG Followed by HyCoSy) | Total
Number analyzed (Participants) | 13 | 6 | 19
Number analyzed (# fallopian tubes) | 26 | 12 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (6.7) | 36.5 (6.7) | 37.3 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Fallopian Tube Patency - HyCoSy vs HSG
Description: Observed flow of fluid/bubbles through fallopian tubes.
Time Frame: At time of procedure
Population: Analysis was per fallopian tube.
Measure: Count of Units; unit: fallopian tubes observed to be closed
Units Other Than Participants: fallopian tubes observed to be closed
Arm/Group | Arm 1 (HyCoSy Followed by HSG) | Arm 2 (HSG Followed by HyCoSy)
Number analyzed (Participants) | 13 | 6
Number analyzed (fallopian tubes observed to be closed) | 26 | 12
fallopian tubes observed to be closed
  Number of tubes closed per first procedure | 24 | 12
  Number of tubes closed per second procedure | 25 | 12
Statistical Analysis 1: Comparison: Arm 1 (HyCoSy Followed by HSG); Test type: Equivalence — Degree of agreement between the 2 Assessors; p < 0.01, Kappa; Degree of agreement / Kappa = 0.48

2. Secondary Outcome: Pain Scores
Description: Patient reported pain scale score on visual pain scale (rated 0 for no pain to 10 for severe pain with corresponding faces)
Time Frame: At time of procedures
Population: Change in patient reported pain scores (pre-procedure minus post-procedure pain scores)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 (HyCoSy Followed by HSG) | Arm 2 (HSG Followed by HyCoSy)
Number analyzed (Participants) | 13 | 6
units on a scale
  HSG post procedure pain score | 1.4 (2.1) | 1.8 (4.0)
  HyCoSy post procedure pain score | 2.4 (3.1) | 2.3 (2.6)
Statistical Analysis 1: Comparison: Arm 1 (HyCoSy Followed by HSG); Test type: Superiority — T-test to determine whether one method had greater reported pain; p < 0.30, t-test, 2 sided; Mean Difference (Final Values) = -0.925, 95% CI 2-sided [-2.69 to 1.00], Standard Deviation 2.71

3. Secondary Outcome: Physician Evaluation of Uterine Cavity
Description: Observed image of uterus (normal or not normal). Assessor commented on uterine cavity to determine whether cavity was normal versus abnormal, e.g., bicornuate uterus or any notable uterine deformity. Data were coded as "normal' or "not normal".
Time Frame: At time of HyCoSy procedure
Population: Number of uteri assessed as 'normal'
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (HyCoSy Followed by HSG) | Arm 2 (HSG Followed by HyCoSy)
Number analyzed (Participants) | 13 | 6
Participants | 13 | 6
Statistical Analysis 1: Comparison: Arm 1 (HyCoSy Followed by HSG); Test type: Superiority; p < 0.67, t-test, 2 sided; Paired t-test (pre-procedure versus post-procedure); Mean Difference (Final Values) = -0.431, 95% CI 2-sided [-2.40 to 1.56], Standard Deviation 2.76

ADVERSE EVENTS:
Time Frame: 1 week after procedures
Groups:
- HyCoSy Followed by HSG: HyCoSy followed by HSG
  HyCoSy: Saline infused sonogram in which air bubbles are delivered via the FemVue saline air device in order to evaluate the patency (openness) of the fallopian tubes
  followed by:
  HSG performed to evaluate the patency (openness) of the fallopian tubes
- Hysterosalpingogram (HSG) Followed by HyCoSy: Hysterosalpingogram (HSG) followed by HyCoSy
  HSG performed to evaluate the patency (openness) of the fallopian tubes
  followed by:
  HyCoSy: Saline infused sonogram in which air bubbles are delivered via the FemVue saline air device in order to evaluate the patency (openness) of the fallopian tubes
Arm/Group | HyCoSy Followed by HSG | Hysterosalpingogram (HSG) Followed by HyCoSy
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/6
Other Adverse Events (participants affected / at risk) | 0/13 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-04-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT02628873/Prot_SAP_ICF_000.pdf